CLINICAL TRIAL: NCT04200937
Title: IT Matters: The Erectile Restoration Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U0670
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- BSC Penile Prothesis Recipients: Men for whom BSC Penile Prothesis is recommended.
  Interventions: Device: Tactra Malleable; Device: Spectra™ Concealable Penile Prothesis; Device: AMS Ambicor™ Inflatable Penile Prosthesis; Device: AMS 700™ Inflatable Penile Prosthesis w/Momentary Squeeze (MS) Pump; Device: AMS 700™ Inflatable Penile Prosthesis w/Tenacio™ Pump

INTERVENTIONS:
Device: Tactra Malleable — The Tactra™ Penile Prosthesis is a sterile, single-use implant that is intended for use in the treatment of chronic, organic, erectile dysfunction (impotence) in adult males who are suitable candidates for implantation procedure.
Device: Spectra™ Concealable Penile Prothesis — The Spectra Penile Prothesis is a sterile, non-pyrogenic, single-use implant that is intended for use in the treatment of chronic, organic, erectile dysfunction (impotence) in men who are determined to be suitable candidates for implantation surgery.
Device: AMS Ambicor™ Inflatable Penile Prosthesis — The AMS Ambicor inflatable penile prothesis intended for use in the treatment of chronic, organic, male erectile dysfunction (impotence) in adult men who are determined to be suitable candidates for implantation surgery.
Device: AMS 700™ Inflatable Penile Prosthesis w/Momentary Squeeze (MS) Pump — The AMS 700 Inflatable Penile Prosthesis is intended for use in the treatment of chronic, organic, male erectile dysfunction (impotence).
Device: AMS 700™ Inflatable Penile Prosthesis w/Tenacio™ Pump — The AMS 700 Inflatable Penile Prosthesis is intended for use in the treatment of chronic, organic, male erectile dysfunction (impotence).

SUMMARY:
The objective of the It MATTERS registry is to collect Real-World Data (RWD) to monitor the safe and effective use of commercially available Boston Scientific Corporation (BSC) penile prostheses

DETAILED DESCRIPTION:
IT MATTERS is a prospective, multicenter, observational registry that is part of planned, active post market clinical follow-up (PMCF) activity associated with each device.

The study will include adult males who undergo penile prothesis implantation with a market approved BSC device to treat erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Males who are determined to be suitable candidates and scheduled to undergo surgical implantation of a market approved BSC penile prothesis by their physician.
3. Willing and able to complete the informed consent process.
4. Willing and able to comply with the follow-up requirements.

Exclusion Criteria:

1. Males who are deemed by their physician as not suitable candidates for a penile prosthesis.
2. In the opinion of the investigator, it is not in best interest of the patient or the study for the patient to participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult males who meet the indications for surgical correction of erectile dysfunction will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to six months in the Erectile Function domain ofthe International Index of Erectile Function (IIEF-EF) questionnaire for Tactra | Baseline to 6 months
  The International Index of Erectile Function (IIEF) is a validated, widely used, multidimensional self-report instrument for the evaluation of erectile function. It consists of 15 items that assess sexual function in five domains: erectile function (Q1, 2, 3, 4, 5,15), orgasmic function (Q9,10), sexual desire (Q11,12), intercourse satisfaction (Q 6,7,8) and overall satisfaction (Q 13,14). A score of 0-5 is awarded to each of the 15 questions. The IIEF-15 total score is the sum of the ordinal responses to the 5 domains.
  The erectile function (EF) domain is the most sensitive domain of the IIEF. IIEF-EF score ranges from 1 to 30 and is derived by scoring 0 (poorest function) to 5 (best function) on each of six questions function (Q1, 2, 3, 4, 5, 15). There are five categories of erectile function based on EF domain score: severe (1-10), moderate (11-16), mild to moderate (17-21), mild (22-25) and no ED (26-30).

SECONDARY OUTCOMES:
Change in depressive symptoms and overall sexual function at Post-Surgery, 6 months, 12 months and annually thereafter post device implantation compared to baseline, as measured by the PHQ-9 Depression Questionnaire and the IIEF: Total Score. | Post-Surgery, 6 months, 12 months and annually thereafter through study completion, an average of 10 years
  The Patient Health Questionnaire (PHQ) is a diagnostic tool for mental health disorders used by health care professionals. The PHQ contains: mood anxiety, alcohol, eating, and somatoform modules. The PHQ-9, is a validated tool specific to depression, scoring each of the 9 DSM-IV criteria. Scored from 0-27, the PHQ-9 is separated into five different diagnoses: minimal depression (0-4), mild depression (5-9), moderate depression (10-14), moderately severe depression (15-19), and severe depression (20-27).
Change in quality of life at 6 months, 12 months, and 24 months post device implantation compared to baseline as measured by the WPAI:GH Questionnaire. | 6 months, 12 months and 24 months
  The WPAI:GH (Work Productivity and Activity Impairment Questionnaire: General Health) is a validated tool that asks a series of questions about the effect of subject health problems, both physical and emotional, on their ability to work and perform regular activities. The WPAI:GH outcomes are expressed as impairment percentages, with higher numbers indicating greater impairment and less productivity, i.e., worse outcomes, as following 6 questions: 1 = currently employed, 2 = hours missed due to health problems, 3 = hours missed other reasons, 4 = hours actually worked, 5 = degree health affected productivity while working, 6 = degree health affected regular activities. Scores are then multiplied by 100 to be expressed in percentages.
Change in erectile function at post-surgery, 12 months and annually post device implantation compared to baseline, as measured by the International Index of Erectile Function Domain (IIEF). | Post-Surgery, 12 months and annually thereafter through study completion, an average of 10 years
  The International Index of Erectile Function (IIEF) is a validated, widely used, multidimensional self-report instrument for the evaluation of erectile function. It consists of 15 items that assess sexual function in five domains: erectile function (Q1, 2, 3, 4, 5,15), orgasmic function (Q9,10), sexual desire (Q11,12), intercourse satisfaction (Q 6,7,8) and overall satisfaction (Q 13,14). A score of 0-5 is awarded to each of the 15 questions. The IIEF-15 total score is the sum of the ordinal responses to the 5 domains.
  The erectile function (EF) domain is the most sensitive domain of the IIEF. IIEF-EF score ranges from 1 to 30 and is derived by scoring 0 (poorest function) to 5 (best function) on each of six questions function (Q1, 2, 3, 4, 5, 15). There are five categories of erectile function based on EF domain score: severe (1-10), moderate (11-16), mild to moderate (17-21), mild (22-25) and no ED (26-30).

OTHER OUTCOMES:
Device satisfaction at post-surgery, 6 months, 12 months and annually thereafter measured by the Likert scale. | Post-surgery, 6 months, 12 months and annually thereafter through study completion, an average of 10 years
  The Likert scale has the options of Very Satisfied, Dissatisfied, Neither Satisfied nor Dissatisfied, Satisfied and Very Satisfied. Responses will be evaluated categorically.
Assess for outcomes and adverse events on AMS Tools at Post Procedure. | Collected only at Post-Procedure
  AMS tools will be assess by a physician survey as part of the post-procedure case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Khera, MD, Principal Investigator — Baylor College of Medicine
Locations (25):
- United States (21):
  - USC Medical Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Tower Urology-Research Facility, Los Angeles, California
  - University of Miami Hospital, Miami, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Willis-Knighton Medical Center, Bossier City, Louisiana
  - Washington University in St. Louis, St Louis, Missouri
  - Duke University Medical Center, Raleigh, North Carolina
  - W.G. Hefner VA Medical Center, Salisbury, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Washington Medical Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- China (3):
  - Peking University First Hospital, Beijing
  - Shanghai General Hospital, Shanghai
  - Shanghai Jiaotong University School of Medicine Renji Hospital, Shanghai
- Johns Hopkins Aramco Healthcare, Dhahran, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No